CLINICAL TRIAL: NCT05714579
Title: Predictive Value of Pre-Transcatheter Aortic Valve Implantation (TAVI) Infrahissian Conduction Time in the Occurrence of Complete Atrioventricular Block in Patients With Preoperative Right Bundle Branch Block
Brief Title: Predictive Value of Pre-TAVI Infrahissian Conduction Time in the Occurrence of Complete Atrioventricular Block
Acronym: TAVHIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor, in consultation with the coordinating investigator, had decided to stop enrolment prematurely because the enrolment rate would not have made it possible to reach the target of 142 patients without increasing the duration of the study
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A02274-39
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- severe aortic stenosis with complete right bundle branch block (Experimental): patients with aortic stenosis undergoing a Transcatheter Aortic Valve Implantation procedure
  Interventions: Procedure: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — The TAVI procedure is performed transfemorally under local anesthesia most often, or more rarely under general anesthesia via the subclavian or transaortic route. Identification is carried out under fluoroscopy in the cardiac catheterization room. The crossing of the aortic valve allows the establishment of a guide at the bottom of the left ventricle. Aortic valve predilation can be performed. The tightness of the device is checked by an aortography. Sometimes, post-dilation of the implanted bioprosthesis proves necessary, particularly in the event of under-deployment or significant para-prosthetic leakage.
  The duration of the intervention is approximately 1 hour.

SUMMARY:
The purpose of the study is implantation of a Pacemaker at 30 days for occurrence of a high-grade conduction disorder per- or post-procedure (yes/no)

DETAILED DESCRIPTION:
The main objective is to assess the predictive value of the pre-TAVI infrahelic conduction time interval (infraheal conduction time measured before percutaneous aortic valve implantation) on the risk of Pacemaker implantation at 30 days post-TAVI, in patients with right bundle branch block prior to surgery.

The aim of the study is to identify a pre-interventional marker of the risk of rhythmological complication after the TAVI procedure (Transcatheter Aortic Valve Implantation), in order to better anticipate it.

This is an interventional, prospective, longitudinal (follow-up: 12 months), multicenter (4 centers) study.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from severe aortic stenosis, eligible for a TAVI procedure (Transcatheter Aortic Valve Implantation) ;
* Patient presenting with complete right bundle branch block during the pre-TAVI electrocardiogram, with QRS interval ≥ 120 ms (depolarization of the ventricles);
* Patient able to understand the information related to the study, to read the information leaflet and agreeing to participate in the study. ;
* Patient having signed a consent.

Exclusion Criteria:

* Contraindication to Transcatheter Aortic Valve Implantation ;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Implantation of a Pacemaker at 30 days | 30 days
  Implantation of a Pacemaker at 30 days for occurrence of a high-grade conduction disorder per- or post-procedure (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Médipôle, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No